CLINICAL TRIAL: NCT03179800
Title: CALM- 2 - Controlling and Lowering Blood Pressure With the MobiusHD™
Acronym: CALM-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Dynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD0447
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Hypertension; Resistant Hypertension
Keywords: Hypertension; Resistant Hypertension; Baroreceptor; BAT
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MobiusHD Implantation (Experimental): MobiusHD Implantation
  Interventions: Device: MobiusHD
- Sham Implantation (Sham Comparator): Sham Implantation
  Interventions: Other: Sham Implantation

INTERVENTIONS:
Device: MobiusHD — The MobiusHD device is a self-expanding nitinol implant that is delivered intravascularly to the internal carotid sinus via the delivery catheter.
  Arms: MobiusHD Implantation
Other: Sham Implantation — Sham Implantation
  Arms: Sham Implantation

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the MobiusHD System in a prospective, randomized, double-blind, sham-controlled multi-center pivotal study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of the MobiusHD System in a prospective, randomized, double-blind, sham-controlled multi-center pivotal study. Patients with resistant hypertension who remain uncontrolled despite pharmacologic treatment with maximum tolerated, guideline-directed anti-hypertensive pharmacologic therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Mean 24 hour ambulatory systolic blood pressure ≥145 mmHg and ≤200 mmHg and stable for at least 8 weeks on a maximally tolerated guideline directed, (JNC8) or their equivalent when those listed are not available dosing regimen consisting of up to 5 antihypertensive medications, with a minimum required dosing regimen of an "A+C+D" antihypertensive medication regimen, where "A" is an angiotensin-converting enzyme Inhibitor or an angiotensin receptor blocker, "C" is a calcium channel blocker, and "D" is a diuretic.

Exclusion Criteria:

* Inadequacy of the carotid anatomy for treatment with the MobiusHD based on carotid angiography.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Change in mean 24-hr sABP from baseline to 180-day | 180-day
  The primary effectiveness endpoint is change in mean 24-hr ambulatory systolic blood pressure (24hr sABP) from baseline to the 180-day visit.

OTHER OUTCOMES:
Safety Assessments - Composite measured at 90-day | 90-day
  Composite measure of death, MI, stroke, device embolization, carotid occlusion, new ipsilateral carotid stenosis requiring surgical or percutaneous intervention, or Bleeding Academic Research Consortium (BARC) 3 or 5 bleeding events as adjudicated by CEC from randomization through the 90-day visit. All adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Williams, MD, Study Chair — University College, London; Gregg Stone, MD, Study Chair — Cardiovascular Research and Education Columbia University Medical Center
Locations (6):
- United States (5):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Southern Illinois University, Springfield, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Carl & Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
- CHU Nancy Centre Coeur et Vaisseaux, Nancy, France

REFERENCES:
- [Derived] Calhoun DA, Schiffrin EL, Flack JM. Resistant Hypertension: An Update. Am J Hypertens. 2019 Jan 1;32(1):1-3. doi: 10.1093/ajh/hpy156. No abstract available. PMID 30407514
- See also: Related Info — http://www.vasculardynamics.com/